CLINICAL TRIAL: NCT00871585
Title: Non-interventional Observational Study to Evaluate Change of PSA Levels in Patients With Advanced Prostate Cancer Treated With Bicalutamide in Combination With Medical or Surgical Castration
Brief Title: Evaluation of Prostate-Specific Antigen (PSA) Levels in Patients With Advanced Prostate Cancer Treated With Bicalutamide
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Ana Marija Gjurovic, Medical&Regulatory Manager, AstraZeneca
Other Study IDs: NIS-OHR-CAS-2008/1
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2010-04-15 (Estimated); Status verified 2010-04

CONDITIONS: Advanced Prostate Cancer
Keywords: bicalutamide; PSA; advanced prostate cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Prospective, non-comparative, non-interventional, observational study to collect and analyse real life environment data on advanced prostate cancer patients receiving combination treatment of medical or surgical castration and bicalutamide according to routine medical practice in Croatia. The main aim is to evaluate change of PSA level and prescribing practices based on prostate cancer stage.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of advanced prostate cancer
* Patients who are already treated with bicalutamide for at least 4 weeks and maximum 12 weeks
* Patients capable of signing ICF

Exclusion Criteria:

* Patients with hypersensitivity to bicalutamide
* Patients on therapy with terfenadin, astemizol or cisapride
* Participation in a clinical study during the last 30 days

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 400 advanced prostate cancer patients (outpatients or hospitalized) treated with bicalutamide in combination with medical or surgical castration according to standard clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2009-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To evaluate change in PSA level following 4-9 months of bicalutamide therapy | PSA - 2 measures (at the time of bicalutamdie introduction and 4-9 m following bicalutamide)

SECONDARY OUTCOMES:
bicalutamide prescribing practice based on prostate cancer stage | 1 measure (at the time of bicalutamde th introduction)
to evaluate PSA level after 4-12 weeks of bicalutamide therapy | PSA - 1 measures (1-3 m following bicalutamide)
to asses time to disease progression based on PSA values | PSA - 3 measures (at the time of bicalutamdie introduction, 1-3 m and 4-9 m following bicalutamide)
to evaluate percentage of patients with disease progression | 2 measures at 1st and 2nd visit
to evaluate withdrawals due to adverse events | 2 measures, at 1st and 2nd visit
to evaluate withdrawals due to Croatian Institute for Health Insurance guidelines for bicalutamide prescription | 2 measures, at 1st and 2nd visit

CONTACTS AND LOCATIONS:
Overall Officials: Ana Marija Gjurovic, Study Director — AstraZeneca; Andreja Hasenohrl, Study Chair — AstraZeneca
Locations (15):
- Croatia (15):
  - Research Site, Čakovec
  - Research Site, Dubrovnik
  - Research Site, Karlovac
  - Research Site, Pula
  - Research Site, Rijeka
  - Research Site, Sisak
  - Research Site, Slavonski Brod
  - Research Site, Split
  - Research Site, Šibenik
  - Research Site, Vinkovci
  - Research Site, Virovitica
  - Research Site, Vukovar
  - Research Site, Zabok
  - Research Site, Zadar
  - Research Site, Zagreb